CLINICAL TRIAL: NCT06559943
Title: The Effect of Kinesio Taping Applications on Pain, Neck Awareness and Functionality in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Yasemin Şahbaz, Dr. Lecturer, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UBeykent-9
Record Dates: First submitted 2024-08-10; First posted 2024-08-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Physiotherapy; Kinesiotape; Chronic Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Physiotherapy + Placebo Kinesio Tape (Placebo Comparator): Following a total of 15 sessions of electro-physical agent treatment, exercise training, 5 days a week for 3 weeks, each session lasting 45 minutes, and traditional physiotherapy 2 days a week for 3 weeks, a total of 6 times applied to the trapezius muscle in the neck area with 0% tension. Kinesiotape will be applied in the form of (I). The tape will be applied twice a week in total, staying for 3 days and leaving one day free after each application.
  Interventions: Other: Traditional Physiotherapy + Placebo Kinesio Tape
- Traditional Physiotherapy + Kinesio Tape Treatment with Inhibition Method (Experimental): Group 2 will receive a total of 15 sessions of electrophysical agent treatment, 45 minutes per session, 5 days a week, for 3 weeks, and kinesiotape treatment with inhibition method in addition to exercise training. Electro-physical agent therapy:
  Intermittent ultrasound at 1.5 w/cm2 for 8 minutes, transcutaneous electrical nerve stimulation, 20 minutes for the trapezius muscle, and hot pack application to the neck area will be applied. Neck isometric exercises, pulley exercise and codman exercise will be applied. Kinesiotape will be applied with the inhibition technique a total of 6 times, following traditional physiotherapy application, 2 days a week for 3 weeks.
  Interventions: Other: Traditional Physiotherapy + Kinesio Tape Treatment with Inhibition Method

INTERVENTIONS:
Other: Traditional Physiotherapy + Placebo Kinesio Tape — Following a total of 15 sessions of electrophysical agent and exercise training, 5 days a week, for 3 weeks, each session lasting 45 minutes, followed by traditional physiotherapy, 2 days a week, for 3 weeks, a total of 6 times, with 0% tension applied to the trapezius muscle in the neck region (I). Kinesiotape will be applied.
  The tape will be applied twice a week in total, staying for 3 days and leaving one day free after each application.
  Arms: Traditional Physiotherapy + Placebo Kinesio Tape
Other: Traditional Physiotherapy + Kinesio Tape Treatment with Inhibition Method — In addition to a total of 15 sessions of electrophysical agents and exercise training, 5 days a week for 3 weeks, each session lasting 45 minutes, kinesio tape will be applied 6 times in total, 2 days a week. Kinesiotape will be cut into an (I) shape (15 cm) with 50% tension and adhered laterally to the C7 joint. In acute cases such as overuse and muscle spasm, it is recommended to apply an inhibition technique that will inhibit the muscle. In the inhibition technique, the direction of the tape should be from the entry point of the muscle to the starting point and the application should be done with very light or light (15 - 25%) tension. In chronic cases, a facilitation technique should be applied to stimulate the weak muscle. The direction of the tape should be from the starting point of the muscle to the attachment point and the application should be done with light or moderate tension (25 - 50%).
  Arms: Traditional Physiotherapy + Kinesio Tape Treatment with Inhibition Method

SUMMARY:
It is important to clarify neck awareness, functional status and pain severity in people with chronic neck pain. Since neck pain, which has become a big problem among the public, cannot be treated definitively, it was aimed to examine the effect of kinesio taping technique on individuals with neck pain. The purpose of the research; To examine the positive and negative effects of kinesio taping applied in addition to traditional treatment on pain, functional status and neck awareness in patients with neck pain. The aim of this study by the researchers is to gain a new perspective on the treatments applied to individuals with neck pain.

DETAILED DESCRIPTION:
Neck pain is a common complaint that can occur for different reasons and is common among the public. The most common musculoskeletal system pathology after low back pain is neck pain. Neck pain symptoms often do not provide a permanent solution. Chronic neck pain is a sensory and emotional experience that affects an individual's quality of life, behavior and professional life. In addition, psychosocial status is also affected due to problems such as health expenses, work attendance problems, and work efficiency. Early diagnosis and identification of risk factors are of great importance to prevent neck pain from turning into a chronic problem. 40-70% of the society complains of neck pain at least once in their lives. About ¼ of these are chronic neck pain. Today, many occupational and personal risk factors for neck pain have been identified. The purpose of the research; The aim of this study is to examine the positive and negative effects of kinesio tape application in addition to traditional treatment on pain, functional status and neck awareness in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in the study and signed the informed consent form,
* Having complained of neck pain for at least 3 months,
* Must be 18 years or older.

Exclusion Criteria:

* Pregnancy
* Loss of function due to neurological or systemic disease,
* Having previously undergone cervical region and spine surgery,
* Having received physiotherapy in the neck and back area in the last 6 months,
* Being on another treatment during the study,
* Having a history of trauma affecting the spine.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 weeks
  Participants will be asked to mark the pain they feel on a 10-centimeter horizontal line. Between 0 and 10, 0 (zero) indicates no pain, while 10 indicates unbearable pain.
Fremantle Neck Awareness Questionnaire | 3 weeks
  Likert type assessing individual-specific altered perception (0 = I never feel like this, 1 = I rarely feel like this, 2 = I feel like this sometimes or some of the time, 3 = I feel like this often, 4 = I feel like this all the time or most of the time) It is a simple survey. The survey asks individuals 9 questions, such as how they perceive their neck in relation to their body and how they perceive their body position. The total score is 0-36 and a high score indicates a poor prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Study Director — Istanbul Beykent University
Locations (1):
- Istanbul Beykent University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Arslanoğlu E, Güzel NA, Çilli B. The Effect of Kinesiotaping Technique on Quadriceps Muscle Strength of Healthy Subjects. Kafkas J Med Sci. 2014;1:23-26. Available from: https://dergipark.org.tr/en/pub/kaftbd/issue/35424/393582.
- [Background] Morris D, Jones D, Ryan H, Ryan CG. The clinical effects of Kinesio(R) Tex taping: A systematic review. Physiother Theory Pract. 2013 May;29(4):259-70. doi: 10.3109/09593985.2012.731675. Epub 2012 Oct 22. PMID 23088702
- [Background] Toprak Celenay S, Mete O, Sari A, Ozer Kaya D. A comparison of kinesio taping and classical massage in addition to cervical stabilization exercise in patients with chronic neck pain. Complement Ther Clin Pract. 2021 May;43:101381. doi: 10.1016/j.ctcp.2021.101381. Epub 2021 Apr 2. PMID 33831805
- [Background] Şimşek Ş, Yağcı N, Oymak Soysal AN, Kaş Özdemir A, Bergin M. Kronik Boyun Ağrısı Olan Bireylerde Ağrı, Fonksiyonel Durum ve Boyun Farkındalığı Arasındaki İlişki. Turk Fizyoter Rehabil Derg. 2022;33(2):106-113. doi: 10.21653/tjpr.979737.